CLINICAL TRIAL: NCT05031871
Title: Pharmacokinetic Study of HR17031 Injection in Healthy Subjects (Single-center, Randomized, Open-label, 4 Cycles, 4 Sequences)
Brief Title: Pharmacokinetics of HR17031 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR17031-102
Record Dates: First submitted 2021-08-16; First posted 2021-09-02 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Experimental): HR17031 injection dose+INS068 injection dose+SHR20004 injection dose+(INS068+SHR20004) injection dose
  Interventions: Drug: HR17031 injection ；INS068 injection；SHR20004 injection
- Treatment group B (Experimental): INS068 injection dose+(INS068+SHR20004)injection dose+ HR17031 injection dose +SHR20004 injection dose
  Interventions: Drug: HR17031 injection ；INS068 injection；SHR20004 injection
- Treatment group C (Experimental): SHR20004 injection dose+ HR17031 injection dose +(INS 068+SHR20004) injection dose+ INS068 injection dose
  Interventions: Drug: HR17031 injection ；INS068 injection；SHR20004 injection
- Treatment group D (Experimental): (INS 068+SHR20004) injection dose+ SHR20004 injection dose+ INS068 injection dose+ HR17031 injection dose
  Interventions: Drug: HR17031 injection ；INS068 injection；SHR20004 injection

INTERVENTIONS:
Drug: HR17031 injection ；INS068 injection；SHR20004 injection — HR17031 injection dose+INS068 injection dose+SHR20004 injection dose+(INS068+SHR20004) injection dose
  Arms: Treatment group A
Drug: HR17031 injection ；INS068 injection；SHR20004 injection — INS068 injection dose+(INS068+SHR20004)injection dose+ HR17031 injection dose +SHR20004 injection dose
  Arms: Treatment group B
Drug: HR17031 injection ；INS068 injection；SHR20004 injection — SHR20004 injection dose+ HR17031 injection dose +(INS 068+SHR20004) injection dose+ INS068 injection dose
  Arms: Treatment group C
Drug: HR17031 injection ；INS068 injection；SHR20004 injection — (INS 068+SHR20004) injection dose+ SHR20004 injection dose+ INS068 injection dose+ HR17031 injection dose
  Arms: Treatment group D

SUMMARY:
To compare the pharmacokinetics and safety of HR17031 injection, SHR20004 injection and/or INS068 injection in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ranges from 18 to 27 kg/m2 (both ends included), and the body weight is ≥50 kg for men and ≥45 kg for women；
2. Fasting blood glucose during the screening is < 6.1 mmol/L；

Exclusion Criteria:

1. It has clinical significance for abnormalities Laboratory examination, if there is a clear reasonable reason, can be retested within a week, with the retest results Whether the subject meets the requirements
2. Severe systemic disease, or a prior history of pancreatitis or other systemic problems within 1 month prior to screening;
3. Participate in any clinical trial of a drug or medical device within 3 months prior to screening (subject to signed informed consent)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Cmax：Maximum observed concentration | Day1 to Day 26
AUC0-t ：Area under the curve from the time of dosing time to the last measurable (positive) concentration； | Day1 to Day 26
AUC0-inf：Area under the curve from time 0 to infinity； | Day1 to Day 26

SECONDARY OUTCOMES:
Tmax ：time of maximum observed concentration | Day1 to Day 26
T1/2：Half-life time ； | Day1 to Day 26
CL/F | Day1 to Day 26
Vz/F | Day1 to Day 26
Serum glucose within 24h after injection | Day1 to Day 23
C-peptide concentrations within 24h after injection | Day1 to Day 23
ADA：anti-drug antibody | Day 1、Day 8、Day15、Day 22 or early termination

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided